CLINICAL TRIAL: NCT01398618
Title: Comparing the Efficacy of Two Preventive Regimens for Adult Household Contacts With Latent Tuberculosis Infection
Brief Title: Comparing Two Preventive Regimens for Latent Tuberculosis Infection (LTBI)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wang, Jann-Yuan/Attending Physician, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201010017M
Record Dates: First submitted 2011-07-01; First posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-06

CONDITIONS: Latent Tuberculosis Infection
Keywords: latent tuberculosis infection; tuberculosis; interferon-gamma release assay; preventive therapy; 9-month isoniazid; 4-month rifampin
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4M-RMP (Experimental): adult household contacts with latent tuberculosis infection receiving 4-month rifampicin preventive therapy
  Interventions: Drug: 4-month rifampin vs. 9-month isoniazid
- 9M-INH (Active Comparator): adult household contact with latent tuberculosis infection receiving 9-month isoniazid preventive therapy
  Interventions: Drug: 4-month rifampin vs. 9-month isoniazid

INTERVENTIONS:
Drug: 4-month rifampin vs. 9-month isoniazid — In the 4M-RMP group, enrolled subjects received 600 mg rifampin daily for 4 months. In the 9M-INH group, enrolled subjects received 300 mg isoniazid daily for 9 months.
  Other Names: 4-month RMP vs. 9-month INH

SUMMARY:
Though still an endemic area, the incidence of tuberculosis (TB) in Taiwan is decreasing in recent years. Further reduction in TB incidence, or even elimination should rely on treatment for LTBI. However, which is the cost-effective screening method or what is the cost-effective regimen in Taiwan is still unclear.

Therefore, the investigators designed this prospective study to follow up adult household contacts with LTBI for 2 years and compare the efficacy of 9-month isoniazid and 4-month rifampicin).

DETAILED DESCRIPTION:
In countries with a low incidence of tuberculosis (TB), most new, active cases have occurred among persons who were once infected, contained this infection, and then later developed active TB. Therefore, identifying persons with latent Mycobacterium tuberculosis infection (LTBI) followed by preventive therapy is an important strategy in public health for TB elimination. Until this decade, the diagnosis of LTBI had been based on contact investigation and tuberculin skin testing (TST). However, false-positive results are not uncommon due to its cross-reactivity with the bacille Calmette-Guérin (BCG) vaccine and some species of non-tuberculosis mycobacteria (NTM), and false-negative results can occur in at least 20% in immunocompromised hosts.

With the application of M. tuberculosis-specific antigens, current interferon-gamma release assays (IGRAs) have been shown to have a better sensitivity and specificity than TST for detecting host response to M. tuberculosis. Therefore, current guidelines for the diagnosis and management of latent tuberculosis infection recommend using IGRA to replace TST. Reports from recent studies comparing the sensitivity, specificity and availability, as well as cost-effective analysis for both tests are inconclusive. The best way varies in different areas, cultures and facilities. Therefore, collecting local data would be very helpful for policy making in public health.

Several regimens have been used in treating LTBI, including 9-month isoniazid, 4-month rifampin, 2-month rifampin plus pyrazinamide, and 3-month isoniazid plus rifampin. Among the 4 regimens, 2-month rifampin plus pyrazinamide has been reported to associate with unacceptable hepatotoxicity and even mortality due to hepatic failure. Therefore, this regimen has now been abandoned in treating LTBI. The treatment completion rate, adverse events, and reduction in risk of developing active TB are similar in 3-month isoniazid plus rifampin as in 6-month Isoniazid. At present, 9-month isoniazid is still the most popular regimen for LTBI, because the toxicity is low, the drug interaction is seldom, and isoniazid has been used for many years. However, the long treatment duration seriously compromises the completion rate. By contrast, rifampin is safe, cheap and more acceptable. Recent studies, including cost-effective analysis, favor using 4-month rifampin in treating LTBI. However, the outcome in these studies is completion rate of preventive therapy, rather than the event of developing active TB. In addition, some use statistic modeling rather conducting a clinical trial.

Though still an endemic area, the incidence of TB in Taiwan is decreasing in recent years. Further reduction in TB incidence, or even elimination should rely on treatment for LTBI. However, which is the cost-effective screening method or what is the cost-effective regimen in Taiwan is still unclear.

Therefore, the investigators designed this prospective study to follow up adult household contacts with LTBI for 2 years and compare the efficacy of 9-month isoniazid and 4-month rifampicin).

ELIGIBILITY:
Inclusion Criteria:

* household contact of patients with newly diagnosed, culture-confirmed pulmonary tuberculosis
* age > 18
* tuberculin skin testing-positive or QuantiFERON-positive
* hemoglobin > 8 g/dL
* neutrophil > 750 /uL
* total bilirubin < 2.5 mg/dL
* aspartic and alanine transaminases < 2 times of upper limit of normal
* willing to receive serology tests for HBV and HCV infection
* no history of allergy to isoniazid and rifampin
* not currently pregnant or breast-feeding

Exclusion Criteria:

* the M. tuberculosis isolate of the index case were isoniazid- or rifampin-resistant
* liver cirrhosis
* clinical or radiographical evidence of active tuberculosis
* active hepatitis
* currently receiving medication that have documented drug interaction with isoniazid or rifampin
* life expectancy < 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants developing active tuberculosis | every 6 months for 2 years

SECONDARY OUTCOMES:
the sensitivity and specificity of tuberculin-skin-testing and QuantiFERON TB-Gold assay for the development of active pulmonary tuberculosis | Every 6 months for 2 years
  Sensitivity: No. of participants who were test-positive among all participants who developed active pulmonary tuberculosis
  Specificity: No. of participants who were test-negative among all participants who did not develop active pulmonary tuberculosis

CONTACTS AND LOCATIONS:
Overall Officials: Jann-Yuan Wang, Ph.D., Principal Investigator — Attending Physician
Locations (2):
- Taiwan (2):
  - Chest Hospital, Department of Health, Executive Yuan, Tainan
  - National Taiwan University Hospital, Taipei

REFERENCES:
- See also: Website of Research Ethic Committee of National Taiwan University Hospital — http://www.ntuh.gov.tw/RECO